CLINICAL TRIAL: NCT04422197
Title: Effect of Botox Injection on Lateral Abdominal Wall Muscles After Major Open Abdominal Surgery
Brief Title: This Randomized Controlled Study Aims to Investigate the Effect of Botox Injection in Abdominal Wall Muscle Post Major Abdominal Surgery in Terms of Postoperative Pain, Incidence of Incisional Hernia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R.19.05.515
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2019-12

CONDITIONS: Hernia, Abdominal
MeSH Terms: conditions — Hernia, Abdominal | interventions — Botulinum Toxins, Type A; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ultrasound-guided botox injection (Active Comparator): Effect of Botox injection on lateral abdominal wall muscles after major open abdominal surgery
  Interventions: Biological: Botox
- Patients with no botox injection (Active Comparator): Patients with major abdominal surgery without botox injection
  Interventions: Procedure: surgery without botox injection

INTERVENTIONS:
Biological: Botox — effect of botox injection in abdominal wall muscle post major abdominal surgery in terms of postoperative pain, incidence of incisional hernia.
  Arms: Patients with ultrasound-guided botox injection
Procedure: surgery without botox injection — surgery without botox injection
  Arms: Patients with no botox injection

SUMMARY:
Aim of the work This randomized controlled study aims to investigate the effect of botox injection in abdominal wall muscle post major abdominal surgery in terms of postoperative pain, incidence of incisional hernia Study design and setting This is a double-blind prospective randomized controlled trial that will be conducted in the general surgery department and colorectal surgery unit of Mansoura University hospital in the period from June 2019 to June2020. The patient's recruitment process will be started and continued for one year after getting the approval from the local Institutional Review Board in Mansoura University in concordance with the Helsinki Declaration Principals. The data will be collected and analyzed prospectively. A signed informed consent will be obtained from every patient before enrollment highlighting the possible future publication. On request, patients can be excluded from the study at any time if they do not want to continue.

ELIGIBILITY:
Inclusion Criteria:

-Patients with major abdominal surgery including trauma and elective exploration surgery, damage control surgery.

Exclusion Criteria:

* pregnancy
* patients with myopathies
* motor polyneuropathies, impaired neuromuscular transmission (Myasthenia Gravis)
* complicated Chronic Obstructive Pulmonary Disease (COPD),
* necrotizing fasciitis of the trunk
* unfit for general anesthesia
* patients with psychiatric disorders
* patients with drug abuse or history of opioid intake
* chronic pain disorder
* coagulopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-02 (Estimated)

PRIMARY OUTCOMES:
incidence of incisional hernia. | one year
  incidence of incisional hernia.Effect of Botox injection on lateral abdominal wall muscles after major open abdominal surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt